CLINICAL TRIAL: NCT04864535
Title: A Pilot Study for the Collection Of Vocalized, Individual Digital Cough Sound Recordings to Screen for COVID-19
Acronym: COVID-Cough
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ResApp Health Limited (Industry)
Collaborators: Strategy Health LLC (Unknown); Ascada Health PC DBA (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21001
Record Dates: First submitted 2021-04-22; First posted 2021-04-29 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-02

CONDITIONS: Covid19
Keywords: COVID-19; Cough
MeSH Terms: conditions — COVID-19; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Recordings of cough sounds from adults — Smartphone recordings of the cough sounds of participants who enrol in the study and obtain a COVID-19 rt-qPCR result.

SUMMARY:
Decentralized clinical study designed to collect cough sounds and self-reported symptoms alongside a COVID-19 realtime quantitative polymerase chain reaction (rt-qPCR) test. The aim of the data collection is to develop a safe and effective cough based digital screening tool for COVID-19.

DETAILED DESCRIPTION:
This study is designed to be administered in a hybrid manner to collect cough sample recordings in association with self-reported symptoms and a COVID-19 rt-qPCR test to investigate whether algorithms can be developed to distinguish COVID-19 positive patients from COVID-19 negative patients using a combination of cough sounds with or without patient-reported symptoms.

Participants will be recruited into two arms with participants entering each arm undergoing the following procedures:

Arm 1 Participants will be recruited into Arm 1 through online marketing campaigns targeted to areas of high COVID-19 incidence as reported by the CDC. Participant recruitment campaign material will direct participants to a Study Landing Page (webpage) (See COVID Cough Study Landing Page - Wire Frame document) that will provide the high-level details of the study including the inclusion/exclusion criteria.

If participants choose to undergo the informed consent process and enroll onto the study, they will download the smartphone-based Study Research App that will virtually perform the following:

* Informed consent completion
* Inclusion/exclusion screening question

If participants are excluded, they will cease to be enrolled on the study (Screen Failure) and the Study Research App will subsequently become inactive. If participants are included, they will proceed within the Study Research App and virtually perform the following:

* Medical symptom questionnaire completion
* Cough sound recording (5 cough sound recordings)
* FDA mandated COVID-19 medical form and participant shipping information After successful completion of the final step presented by the Study Research App, participants will be shipped via FedEx a 2-day shipping FDA EUA authorized at-home self-administered, saliva-based COVID-19 rt-qPCR test developed and analyzed by a CLIA, CAP, and NYS DOH certified laboratory in Secaucus, NJ.

Participants will receive their COVID-19 rt-qPCR test within a test kit box that will also contain a study flyer designed to prompt the participant to reengage the Study Research App. Participants will also be prompted by an email sent out at the time of delivery of their COVID-19 test kit. If during the study assessment of the data shows that participant retention is poor the study PI may implement a single SMS set to the participant at the time of delivery to add an extra reminder to perform the following steps within the Study Research App alongside performing their self-administered COVID-19 test:

* Medical symptom questionnaire completion
* Cough sound recording (5 cough sound recordings) Participants will be provided a pre-paid FedEx shipping label with which to return their COVID-19 test to the study partner laboratory which will analyze tests and report test results to participants as per their standard operating procedures.

Data collected by the Study Research App will be encrypted locally on the participant's phone and uploaded to a secure, restricted access, HIPAA compliant ShareFile folder.

Data collected by the Study Research App and partner lab will also be recorded in an electronic Clinical Data Management system for security and data privacy (See COVID Cough Study Case Report Form Document).

Arm 2 Potential participants will be identified by the study staff at a partner testing site ("Partner Site") based on recently (<24 hours) receiving a positive COVID-19 test result on Rapid PCR testing. Eligible participants will be called back to attend the Partner Site within <48 hours of undergoing their COVID-19 test.

Eligible subjects will be consented and enrolled into the study through a paper Informed Consent Form that is signed in person at the Partner Site.

After enrollment, participants will be asked questions regarding any signs and symptoms of respiratory disease after which the enrolled subject's cough sounds will be captured (5 cough sounds are required) using the COVID Cough In-clinic Study application software installed on a study smartphone utilized by the Partner Site study staff. The COVID Cough In-clinic Study application software is a piece of software that mimics the cough recording capture elements of the Study Research App and provides the ability to enter a subject's date of birth for file identification purposes.

As this is an observational study, after cough recording capture the Partner Site study staff will only receive a unique cough recording identifier by the study smartphone which will be recorded in the participant's eCRF.

In both study arms participants will receive a copy of their completed ICF upon completing the ICF process.

ELIGIBILITY:
Inclusion Criteria:

* be aged 21 years and older;
* be a resident of the USA;
* have a personal (i.e., not shared) iPhone 6s or newer running iOS 14 or later;
* be able to read and understand English;
* be able to provide informed consent;
* be able to provide at least 5 coughs (voluntary and/or spontaneous);
* if enrolling online in Arm 1, the participant must be unvaccinated against COVID-19 (have not received one or more doses of a COVID-19 vaccine at any time before study enrolment)

Exclusion Criteria:

* have one or more medical contraindication to voluntary cough, including the following:

  * Severe respiratory distress;
  * History of pneumothorax;
  * Eye, chest, or abdominal surgery within 3 months of enrolling for the study; or
  * Hemoptysis (coughing up of blood) within 1 month of enrolling for the study;

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 100 participants who test positive for COVID-19 on rt-qPCR will be recruited. Based on average COVID-19 incidence rates in high incidence US geographies (~8-12%), this study will enrol a cohort of up to 1500 participants on a rolling basis, to allow for sufficient cough recordings from COVID-19 positive participants to be collected for analysis.
  Participants will be aged 21 years and older and will not be excluded based on gender, demographic group, or geographic location within the US.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Collection of cough sound recordings and self-reported symptoms from a minimum of 100 COVID-19 positive participants as identified by rt-qPCR. | 3 months
  Cough sound recordings and symptoms from COVID-positive patients
Development of an algorithm that uses a combination of cough sounds and self-reported symptoms that is capable of distinguishing between COVID-19 positive and COVID-19 negative participants. | 3 months
  Cough sound algorithm that distinguishes with COVID-19 positive and negative cough sounds.

SECONDARY OUTCOMES:
Development of an algorithm that uses cough sounds that is capable of distinguishing between COVID-19 positive and COVID-19 negative participants. | 3 months
  Algorithm for software application to distinguish between COVID-19 positive and negative coughs

OTHER OUTCOMES:
Development of an algorithm that uses a combination of cough sounds and patient-reported symptoms that is capable of predicting rt-qPCR Ct value for a participant. | 3 months
  Algorithm could predict similar result to a rt-qPCR Ct value

CONTACTS AND LOCATIONS:
Overall Officials: Shrawan Patel, MBBS BSc, Principal Investigator — Strategy Health LLC
Locations (1):
- Strategy Health LLC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No